CLINICAL TRIAL: NCT00089687
Title: GBR 12909 Study in Cocaine Experienced African American Volunteers
Brief Title: GBR 12909 Study in Cocaine Experienced African American Volunteers - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CPU-0005-1
Record Dates: First submitted 2004-08-10; First posted 2004-08-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-01

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — vanoxerine

INTERVENTIONS:
Drug: GBR 12909

SUMMARY:
The purpose of this study is to assess GBR 12909 in cocaine experienced African American Volunteers.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled, safety and pharmacology study with 75 mg dosage of GBR 12909 in cocaine experienced African American Volunteers. Particular interest is being given to the hematological safety data.

ELIGIBILITY:
Inclusion Criteria:

* Must be within 20% of ideal body weight and must weigh at least 45 kg.
* Must understand the study procedures and provide written informed consent.
* Must meet DSM-4 criteria for abuse or dependence on cocaine.
* Must be non-treatment seeking at the time of the study.

Exclusion Criteria:

* Please contact the study site for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2004-04; Study Completion 2005-05

PRIMARY OUTCOMES:
pharmacokinetic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States